CLINICAL TRIAL: NCT05577715
Title: A Phase 2, Open-label, Randomized Study of MORAb-202 (Farletuzumab Ecteribulin), a Folate Receptor Alpha-targeting Antibody-Drug Conjugate, in Participants With Metastatic Non-Small Cell Lung Cancer (NSCLC) Adenocarcinoma (AC) After Progression on Prior Therapies
Brief Title: A Study of MORAb-202 in Participants With Previously Treated Metastatic Non-Small Cell Lung Cancer (NSCLC) Adenocarcinoma (AC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA116-003; 2022-000131-23 (EudraCT Number); MORAb-202-G000-203 (Other: Eisai Protocol Number)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; MORAb-202; Farletuzumab ecteribulin; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — MORAb-202

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MORAb-202 (Experimental)
  Interventions: Drug: MORAb-202

INTERVENTIONS:
Drug: MORAb-202 — Specified dose on specified days
  Other Names: Farletuzumab Ecteribulin; BMS-986445

SUMMARY:
The aim of this study is to characterize the safety and tolerability of MORAb-202, and to assess the objective response rate in participants with previously treated, metastatic NSCLC AC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented metastatic NSCLC AC (as defined by the 8th International Association for the Study of Lung Cancer Classification).
* Measurable target disease assessed by the investigator according to RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1

Exclusion Criteria:

* NSCLC histologies other than AC (ie, squamous cell carcinoma, large cell carcinoma).
* Significant third-space fluid retention (eg, ascites or pleural effusion) that requires repeated drainage.
* Prior pneumonectomy. Prior lobectomy and segmentectomy are allowed > 12 months before treatment.
* Recent chest radiotherapy. Participants with chest or chest wall radiation may be permitted if chest radiation is documented > 6 months before starting study treatment.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (13):
  - Local Institution - 0007, Orange, California
  - Local Institution - 0035, Lone Tree, Colorado
  - Local Institution - 0043, Clermont, Florida
  - Local Institution - 0010, Orange City, Florida
  - Local Institution - 0001, Marietta, Georgia
  - Local Institution - 0005, Louisville, Kentucky
  - Local Institution - 0044, Silver Spring, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Local Institution - 0002, Kansas City, Missouri
  - Local Institution - 0011, Charlotte, North Carolina
  - Local Institution - 0034, Arlington, Texas
  - Local Institution - 0045, Flower Mound, Texas
  - Local Institution - 0033, Fairfax, Virginia
- Australia (3):
  - Local Institution - 0040, Wollongong, NS
  - Local Institution - 0012, Ballarat Central, Victoria
  - Local Institution - 0022, Murdoch, Western Australia
- Belgium (2):
  - Local Institution - 0039, Mons, WHT
  - Local Institution - 0036, Roeselare
- Chile (4):
  - Local Institution - 0028, Providencia, SA
  - Local Institution - 0030, Independencia
  - Local Institution - 0027, Recoleta
  - Local Institution - 0023, Santiago
- France (4):
  - Local Institution - 0017, Rouen
  - Local Institution - 0015, Suresnes
  - Local Institution - 0014, Toulon
  - Local Institution - 0038, Villejuif
- Spain (7):
  - Local Institution - 0020, Málaga, MA
  - Local Institution - 0019, Majadahonda (Madrid), M
  - Local Institution - 0025, Barcelona
  - Local Institution - 0021, Barcelona
  - Local Institution - 0018, Madrid
  - Local Institution - 0026, Santiago de Compostela
  - Local Institution - 0031, Seville

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- MORAb-202 25mg/m^2: Participants with metastatic non-small cell lung cancer (NSCLC) adenocarcinoma after progression on prior therapies received 25mg/m^2 intravenous infusion once every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | MORAb-202 25mg/m^2
Started | 31
Completed | 7
Not Completed | 24
Not completed — Withdrawal by Subject | 1
Not completed — STUDY TERMINATED BY SPONSOR | 16
Not completed — Lost to Follow-up | 1
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | MORAb-202 25mg/m^2
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 30

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Per Investigator
Description: ORR is defined as the percentage of participants whose best overall response (BOR) is either CR or PR per response evaluation criteria in solid tumors (RECIST) v1.1 based on Clopper-Pearson method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of randomization to the date of first objectively documented progression or death, whichever occurs first (Up to approximately 12 months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MORAb-202 25mg/m^2
Number analyzed (Participants) | 31
percentage of participants | 9.7 [2.0 to 25.8]

2. Primary Outcome: Number of Participants With Drug -Related Adverse Events Leading to Discontinuation
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 12 months).
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 25mg/m^2
Number analyzed (Participants) | 31
Participants | 3

3. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events and Adverse Event of Special Interest (AESI) and Deaths and Grade 3/4 Laboratory Abnormalities (SI Units)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Serious adverse events (SAE) are defined as any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death).
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 12 months).
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 25mg/m^2
Number analyzed (Participants) | 31
Participants
  Adverse Events Grade 1 | 10
  Adverse Events Grade 2 | 5
  Adverse Events Grade 3 | 3
  Adverse Events Grade 4 | 0
  Adverse Events Grade 5 | 0
  Serious Adverse Events (Any Grade) | 7
  Serious Adverse Events (Grade 3/4) | 7
  Serious Adverse Events Grade 5 | 1
  Drug related SAEs Any Grade | 2
  Drug related SAEs Grade 3-4 | 2
  Drug related SAEs Grade 5 | 0
  Drug related AEs Grade 1 | 10
  Drug related AEs Grade 2 | 5
  Drug related AEs Grade 3 | 3
  Drug related AEs Grade 4 | 0
  Drug related AEs Grade 5 | 0
  AESI - Pneumonitis | 2
  AESI - Bronchospasm | 1
  Infusion related reaction | 1
  Deaths | 7
  Lymphocytes (ABSOLUTE) Grade 3 | 1
  Creatinine - Grade 3 | 2

4. Secondary Outcome: Disease Control Rate as Per Investigator
Description: Disease Control Rate (DCR) is defined as the number of randomized participants who achieve a BOR of confirmed CR, confirmed PR, or stable disease (SD) divided by the number of all randomized participants. per response evaluation criteria in solid tumors (RECIST) v1.1 based on Clopper-Pearson method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MORAb-202 25mg/m^2
Number analyzed (Participants) | 31
percentage of participants | 67.7 [48.6 to 83.3]

5. Secondary Outcome: Duration of Response as Per Investigator
Description: DOR for a participant with a best overall response (BOR) of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death, whichever occurs first.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: All Randomized Participants. Only responders (CR or PR) were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | MORAb-202 25mg/m^2
Number analyzed (Participants) | 3
months | NA [NA to NA] — Not estimated due to insufficient number of events.

6. Secondary Outcome: Progression Free-Survival as Per Investigator
Description: PFS is defined for all randomized participants as the date from randomization to the date of the documentation of disease progression or death due to any cause, whichever is earlier.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: as for outcome 1
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MORAb-202 25mg/m^2
Number analyzed (Participants) | 31
months | 3.52 [2.60 to 5.42]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and non-serious adverse events were collected from first dose until 30 days after last dose (Up to approximately 12 months).
Arm/Group | MORAb-202 25mg/m^2
All-Cause Mortality (participants affected / at risk) | 7/31
Serious Adverse Events (participants affected / at risk) | 7/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-202 25mg/m^2 (N=31)
Hip fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-202 25mg/m^2 (N=31)
Anaemia (Blood and lymphatic system disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 6
Fatigue (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 3
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Proteinuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT05577715/Prot_SAP_000.pdf